CLINICAL TRIAL: NCT05022147
Title: ENGAGE-PD: Enhancing Gait Using Alternating-Frequency DBS in Parkinson Disease
Brief Title: Enhancing Gait Using Alternating-Frequency DBS in Parkinson Disease
Acronym: ENGAGE-PD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: James Liao (Other)
Responsible Party: Sponsor-Investigator, James Liao, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-739
Record Dates: First submitted 2021-08-09; First posted 2021-08-26 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic; Disease Progression; Subthalamic Nucleus; Accidental Fall; Deep Brain Stimulation
Keywords: Postural Instability; Gait Impairment; Freezing of Gait; DBS; Frequency; Low; Alternating; Variable; High
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic; Disease Progression

STUDY DESIGN:
Intervention Model Description: On a single day, participants will switch between six DBS frequency conditions. Gait and body kinematics will be monitored during these conditions. The order that participants experience the six conditions will be randomized, and participants will be blinded to the condition. In addition, the assessments will be performed OFF and then repeated ON medication.
Masking Description: There is only one arm in the study. Participants will be masked to which device intervention is active, but they will not be masked to the medication state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Alternating-Frequency DBS (Experimental): In this single-arm study, all participants will receive all interventions in a crossover fashion.
  Interventions: Device: High-Frequency-Only Stimulation; Device: Low-Frequency-Only Stimulation; Device: Alternating, 50 sec High-Frequency, 10 sec Low-Frequency Stimulation; Device: Alternating, 50 sec High-Frequency, 50 sec Low-Frequency Stimulation; Device: Alternating, 10 sec High-Frequency, 50 sec Low-Frequency Stimulation; Device: Alternating, 10 sec High-Frequency, 10 sec Low-Frequency Stimulation; Drug: OFF Dopaminergic Medication; Drug: ON Dopaminergic Medication

INTERVENTIONS:
Device: High-Frequency-Only Stimulation — Control condition, constant high-frequency DBS stimulation (130Hz)
Device: Low-Frequency-Only Stimulation — Experimental condition, constant low-frequency DBS stimulation (60 Hz)
Device: Alternating, 50 sec High-Frequency, 10 sec Low-Frequency Stimulation — Experimental condition where stimulation frequency is changed from high (130Hz) to low (60Hz) frequency. The time interval for each frequency is 50 seconds for high, and 10 seconds for low, respectively.
Device: Alternating, 50 sec High-Frequency, 50 sec Low-Frequency Stimulation — Experimental condition where stimulation frequency is changed from high (130Hz) to low (60Hz) frequency. The time interval for each frequency is 50 seconds for high, and 50 seconds for low, respectively.
Device: Alternating, 10 sec High-Frequency, 50 sec Low-Frequency Stimulation — Experimental condition where stimulation frequency is changed from high (130Hz) to low (60Hz) frequency. The time interval for each frequency is 10 seconds for high, and 50 seconds for low, respectively.
Device: Alternating, 10 sec High-Frequency, 10 sec Low-Frequency Stimulation — Experimental condition where stimulation frequency is changed from high (130Hz) to low (60Hz) frequency. The time interval for each frequency is 10 seconds for high, and 10 seconds for low, respectively.
Drug: OFF Dopaminergic Medication — All six device interventions will be performed in medication OFF state
Drug: ON Dopaminergic Medication — All six device interventions will be performed in medication ON state

SUMMARY:
The purpose of this study is to assess how alternating-frequency Deep Brain Stimulation (DBS) works to improve postural instability and gait, while also treating other motor symptoms of Parkinson Disease (PD).

DETAILED DESCRIPTION:
Postural instability, gait impairment, and falls are among the greatest unmet needs in Parkinson disease (PD). A single fall can be catastrophic, and impairments that limit mobility lead to social isolation or depression, and adversely affect bone and cardiovascular health. Unfortunately, postural instability and gait disorders are refractory to current pharmacological and surgical treatments, including deep brain stimulation (DBS). This project will directly address this pressing need. We will recruit participants to perform a gait task, using a new, alternating DBS frequency paradigm, while body movements and neural signals are recorded. The findings will lead to improved therapies to address these symptoms in the future.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral STN DBS for PD
* Medtronic Percept PC implanted DBS battery/pulse generator/recording system
* Presence of balance and/or walking impairment and/or freezing of gait
* Can walk without assistance, OFF meds, based on yes/no verbal response

Exclusion Criteria:

* Severity of gait impairment should not require dependency to walker or cane
* Cannot tolerate monopolar stimulation at either of the two middle electrode contacts (prerequisite for the recording mode of the DBS) at high frequency (130 Hz) or low frequency (60 Hz).
* Concomitant conditions that may affect significantly the evaluation of balance or gait, including orthopedic, rheumatologic or other neurological diseases
* Contraindication to physical therapy
* Age < 21
* Diagnosis of dementia
* Not agreeable to having video taken of entire research visit

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Stride Time Coefficient of Variation | During the intervention
  Marker of gait instability, derived from kinematic recordings from body-worn wireless sensors.
Percentage of Time with Tremor Present | During the intervention
  Marker of tremor severity, derived from kinematic recordings from body-worn wireless sensors.
Tremor Amplitude | During the intervention
  Marker of tremor severity, derived from kinematic recordings from body-worn wireless sensors.

SECONDARY OUTCOMES:
Total Freezing Time | During the intervention
  Marker of gait instability, derived from kinematic recordings from body-worn wireless sensors.
Freezing Index | During the intervention
  Marker of gait instability, derived from kinematic recordings from body-worn wireless sensors.
Gait Velocity | During the intervention
  Marker of bradykinesia, derived from kinematic recordings from body-worn wireless sensors.
Step Cadence | During the intervention
  Marker of bradykinesia, derived from kinematic recordings from body-worn wireless sensors.
LFP and EEG power spectrum correlation with behavior and kinematics | During the intervention
  Neural recordings (LFP = Local Field Potential and EEG = Electroencephalogram) from the DBS electrode and from EEG electrodes will be analyzed in the frequency domain. Assessed frequency bands will include delta, theta, alpha, beta, and gamma activity. These will be correlated with behavior and kinematic recordings to determine the neural correlates of gait instability and other parkinsonian symptoms.
LFP and EEG connectivity correlation with behavior and kinematics | During the intervention
  Neural recordings (LFP = Local Field Potential and EEG = Electroencephalogram) consist of multiple channels of simultaneously measured electrical activity. Connectivity is a measure of correlations between each pair of recorded and postprocessed channels, at each frequency band, over time. A machine learning algorithm will be trained to correlate the connectivity to behavior and kinematic recordings, to determine the neural correlates of gait instability and other parkinsonian symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: James Liao, MD PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
At time of publication, a point of contact individual on the study team will be identified. Third parties will be able to request access to de-identified data used to support the publication findings by application to the Cleveland Clinic IRB. A data use agreement will be put in place between the CCF Cleveland Clinic and this third party for approved use of the data.